CLINICAL TRIAL: NCT02263248
Title: Incomplete Response in Late-Life Depression: Getting to Remission With Buprenorphine
Acronym: (IRLGREY-B)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Reckitt Benckiser LLC (Industry)
Responsible Party: Principal Investigator, Daniel Blumberger, Dr. Daniel. M. Blumberger, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 035/2014
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Venlafaxine Hydrochloride; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- venlafaxine XR plus buprenorphine (Experimental): Drug Intervention: venlafaxine XR plus buprenorphine Dosage varies. Subject remains on antidepressant throughout the 32 week study. Will be randomized to buprenorphine or placebo for up to 16 weeks.
  Interventions: Drug: venlafaxine; Drug: buprenorphine
- venlafaxine XR plus placebo (Placebo Comparator): Drug Intervention: venlafaxine XR plus placebo Dosage varies . Subject remains on antidepressant throughout the 32 weeks study. Will be randomized to buprenorphine or placebo for up to 16 weeks
  Interventions: Drug: venlafaxine; Drug: placebo

INTERVENTIONS:
Drug: venlafaxine — slow titration to a maximum of 300 mg per day. will remain on venlafaxine XR for upto 32 weeks.
  Other Names: Effexor
Drug: buprenorphine — randomized to either buprenorphine or placebo, dose range from 0.2 mg qd/ to 1.2 mg qd
  Other Names: Temgesic; Subutex; Suboxone
  Arms: venlafaxine XR plus buprenorphine
Drug: placebo — patients will remain on venlafaxine XR and be randomzied to receive either placebo or buprenorphine for 8 weeks. at the end of 8 weeks those who did not receive buprenorphine will be given an opportunity to try it.
  Arms: venlafaxine XR plus placebo

SUMMARY:
The Investigators are conducting a research study to learn about the safety and benefit of using a medication called buprenorphine for patient with difficult to treat depression . This research study is testing whether combining two medications will be effective in treating depression when initial treatment with just one antidepressant does not relieve the depressive symptoms ; this is what is called " difficult to treat depression " or " treatment resistant depression ". The two medication the investigators are using are " an anti-depressant medication called venlafaxine XR ( the generic form of Effexor ) and buprenorphine . Buprenorphine is a medication that is FDA approved for the treatment of opioid dependence. The investigators are testing whether adding buprenorphine to venlafaxine enhances treatment response.

DETAILED DESCRIPTION:
The aim of this study is to examine the feasibility, safety, and tolerability of buprenorphine (BPN) as a novel treatment for late-life treatment resistant depression (LL-TRD). The investigators aim to use a clinical trial methodology common to all three sites, and to examine the mechanism of action (MOA) of BPN using translational neuroscience methods. Over ½ of seniors with depression fail to respond to traditional antidepressants.19,20 Modulation of the opiate system with BPN offers a novel mechanistic approach to improve the lives of patients with LL-TRD, with a safety profile potentially superior to current augmentation strategies such as antipsychotics, lithium, ECT, and surgical interventions (e.g., deep brain or vagal nerve stimulation).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Major depressive disorder (MDD), single or recurrent, as diagnosed by the SCID-IV (or SCID-5 if available)
3. MADRS > 15
4. Has or agrees to establish a clinical relationship with primary care physician (PCP).
5. Availability of an informant (e.g., emergency contact) is encouraged but not required for study participation

Exclusion Criteria:

1. Inability to provide informed consent
2. Depressive symptoms not severe enough (i.e., MADRS < 15) at the baseline assessments
3. Dementia, as defined by 3MS < 80 and clinical evidence of dementia
4. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms, as diagnosed by the SCID
5. Abuse of or dependence on alcohol or other substances within the past 3 months as determined by SCID, and score of > 8 on AUDIT-C and confirmed by study physician interview
6. High risk for suicide (e.g., active SI and/or current/recent intent or plan) AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases
7. Contraindication to venlafaxine or buprenorphine as determined by PCP and study physician including history of intolerance of either venlafaxine or buprenorphine in the study target dosage range (venlafaxine at up to 300 mg/day; buprenorphine at up to 1.2 mg/day)
8. Inability to communicate in English (i.e., interview cannot be conducted without an interpreter; subject largely unable to understand questions and cannot respond in English)
9. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
10. Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management. This will be determined based on information from the patient's personal physician and study physician's clinical judgment. Referral to the patient's personal physician or to a general practitioner will be made in these cases
11. Subjects taking psychotropic medications that cannot be safely tapered and discontinued prior to study initiation. The following exceptions are allowed if they have been taken at a stable dose for at least 4 weeks prior to study entry and there is not a plan to change the dose during the next 32 -36 weeks: benzodiazepines up to 2 mg/d lorazepam equivalent; other sedative-hypnotics (e.g., zolpidem, zaleplon, eszopiclone); gabapentin if prescribed for non-psychiatric indication (e.g., neuropathy)
12. History of opiate abuse or dependence
13. Severe pain, defined as > 7 on 0-10 numeric rating scale for pain
14. Concomitant use of strong or moderate CYP3A4 inhibitor (indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketonazole, nefazodone, saquinovir, telithromycin, aprepitant, erythromycin, fluconazole, grapefruit juice, verapamil, diltiazem)
15. Refusal to stop all opioids (to avoid precipitating opioid withdrawal)
16. Refusal to discontinue all alcohol (to reduce the risk of respiratory depression)
17. Hepatic impairment (AST/ALT > 1.5 times upper normal)
18. Estimated Glomerular Filtration Rate (GFR) < 20 ml/min
19. Inability/refusal to identify a person as an emergency contact

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-19 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
The Montgomery-Asberg Depression Rating Scale | 32 weeks
  MADRS at baseline will establish study eligibility and will assess treatment-sensitive change in MDD.

SECONDARY OUTCOMES:
Suicidal Ideation Scale ( SIS) | 32 weeks
  Assess suicidal ideation and previous suicide attempts
Brief Symptom Inventory for Anxiety | 32 weeks
Numeric Scale of Pain ( NRS-P) | 16 weeks
Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) | 16 weeks
  Assess overall burden or degree of interference in day-to-day activities and function due to the side effects attributable specifically to the antidepressant (in this case, buprenorphine) treatment
Antidepressant Side Effect Checklist (ASEC) | 16 weeks
  Assessment of side- effects

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Blumberger, MD, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buchalter ELF, Oughli HA, Lenze EJ, Dixon D, Miller JP, Blumberger DM, Karp JF, Reynolds CF 3rd, Mulsant BH. Predicting Remission in Late-Life Major Depression: A Clinical Algorithm Based Upon Past Treatment History. J Clin Psychiatry. 2019 Dec 10;80(6):18m12483. doi: 10.4088/JCP.18m12483. PMID 31846575